CLINICAL TRIAL: NCT03844724
Title: Safety and Efficacy of ZENFlow™ Drug-eluting PTA Balloon Dilatation Catheter in the Treatment of Iliac, Femoral and Popliteal Artery Stenosis or Occlusion
Brief Title: Drug-eluting PTA Balloon Dilatation Catheter in the Treatment of Peripheral Artery Stenosis or Occlusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Zylox Medical Device Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZYLOX2014001
Record Dates: First submitted 2019-02-13; First posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Peripheral Arterial Disease; Iliac Artery Stenosis; Femoral Artery Stenosis; Popliteal Artery Stenosis; Iliac Artery Occlusion; Femoral Artery Occlusion; Popliteal Artery Occlusion
Keywords: Peripheral Arterial Disease; Drug-eluting PTA Balloon Dilatation Catheter; Late Lumen Loss（6 months）
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): subjects using the drug-eluting PTA balloon dilatation catheter
  Interventions: Device: ZENFlow™ Drug-eluting PTA Balloon Dilatation Catheter
- Group B (Active Comparator): subjects using the peripheral balloon dilatation catheter
  Interventions: Device: Peripheral Balloon Dilatation Catheter

INTERVENTIONS:
Device: ZENFlow™ Drug-eluting PTA Balloon Dilatation Catheter — Digital subtraction angiography（DSA）
  Arms: Group A
Device: Peripheral Balloon Dilatation Catheter — Digital subtraction angiography（DSA）
  Arms: Group B

SUMMARY:
Clinical study on safety and efficacy of ZENFlow™ drug-eluting PTA balloon dilatation catheter in the treatment of iliac, femoral and popliteal artery stenosis or occlusion

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the safety and efficacy of ZENFlow™ drug-eluting PTA balloon dilatation catheter (paclitaxel 3±1 μg/mm2 balloon surface area) in the treatment of iliac artery, femoral artery and popliteal stenosis or occlusive lesions compared with conventional PTA balloon dilatation catheter.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 85 years old, male or female
* Subject's target lesions were stenosis and/or occlusion
* Subjects were able to understand the purpose of the study, demonstrate full compliance with the program and sign informed consent

Exclusion Criteria:

* Pregnant woman or who's pregnancy test is positive
* Lactation period woman or woman/man with fertility plan

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2015-04-10 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
Late Lumen Loss at 6 months after operation | 6 months
  Late Lumen Loss

SECONDARY OUTCOMES:
The incidence of major adverse events | 12 months
  Related to death of clinical trials
Adverse Event | Preoperative、Intraoperative、up to 1 month、3 months、6 months、9 months、12 months
  Adverse medical events, whether or not related to the medical device

CONTACTS AND LOCATIONS:
Overall Officials: Changwei Liu, Principal Investigator — Peking Union Medical College Hospital

REFERENCES:
- [Derived] Ni L, Ye W, Zhang L, Jin X, Shu C, Jiang JS, Yang M, Wu DM, Li M, Yu GF, Yang J, Huang JH, Wang XB, Li XQ, Jiang WL, Wu ZQ, Liu CW. A Multicenter Randomized Trial Assessing ZENFlow Carrier-Free Drug-Coated Balloon for the Treatment of Femoropopliteal Artery Lesions. Front Cardiovasc Med. 2022 Mar 15;9:821672. doi: 10.3389/fcvm.2022.821672. eCollection 2022. PMID 35391838